CLINICAL TRIAL: NCT05561023
Title: Phase Ⅰa Clinical Study of Hawthorn Red Pigment Combined With Standard Analgesic for Refractory Cancer Pain
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HBG-01/SYLT-024
Record Dates: First submitted 2022-09-12; First posted 2022-09-30 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Hawthorn Red Combined Refractory Cancer Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Phase Ⅰ a clinical study (Other): "3 + 3" dose escalation scheme
  Interventions: Drug: Hawthorn red pigment

INTERVENTIONS:
Drug: Hawthorn red pigment — For patients with refractory cancer pain who meet the enrollment conditions, on the basis of the clinician's normal adjustment of the analgesic regimen (the initial adjustment is the first day), the dose ramp up study of Hawthorn red pigment was started on the third day. The Hawthorn red dose group includes 10 tablets → 15 tablets → 20 tablets / time, orally, twice a day.
  "3 + 3" dose escalation scheme

SUMMARY:
To evaluate the safety and tolerance of Hawthorn red pigment in the treatment of cancer pain

Determine the maximum tolerated dose (MTD, if any) of Hawthorn red pigment and the recommended dose for phase II clinical study (RP2D)

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-80 years with malignant tumor confirmed by pathology;
2. Refractory cancer pain, that is, patients coexist: 1) digital score of persistent pain ≥ 4 points and / or number of eruptive pain ≥ 3 times / day; 2) Following the relevant guidelines for cancer pain treatment, the pain relief of patients treated with opioids alone and / or combined with adjuvant analgesics for 1-2 weeks is still unsatisfactory and / or intolerable adverse reactions occur;
3. Patients who need chemotherapy, long-term hormone, targeted therapy or bisphosphate therapy had stable anti-tumor therapy before randomization;
4. Patients or their nursing staff can fill in the survey form;
5. Correctly understand and cooperate with medical staff in medication guidance;
6. No mental illness;
7. ECOG-ps ≤ 3 points; 8) Did not participate in the drug test (including the test drug) within one month before the test;
8. The subjects volunteered and signed the informed consent.

Exclusion Criteria:

1. patient is diagnosed with non cancerous pain or pain of unknown cause;
2. Postoperative pain of patients;
3. Patients with paralytic intestinal obstruction;
4. Patients with metastatic brain cancer;
5. Patients with opioid allergy / addiction;
6. Abnormal laboratory results with obvious clinical significance, such as creatinine ≥ upper limit of normal value, ALT or AST ≥ 2.5 times of upper limit of normal value (liver metastasis patients or primary liver cancer ≥ 5 times of upper limit of normal value), or child C level of liver function;
7. Patients who cannot take drugs orally;
8. Uncontrollable nausea and vomiting;
9. Patients with a history of gastritis and gastric ulcer;
10. Patients who need to use nonsteroidal drugs and steroid hormone drugs for analgesia;
11. Diabetes patients who can't control blood sugar stably;
12. Pregnant and lactating women; Subjects with pregnancy plans within 1 month after the trial (including male subjects);
13. Alcoholics;
14. Patients with cognitive impairment;
15. Patients with severe depression;
16. Diseases and conditions that other researchers consider not to be included.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
AE, SAE and DLT, MTD (if any), RP2D | 1 month
  Occurrence and frequency of AE, SAE and DLT, MTD (if any), RP2D, Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

SECONDARY OUTCOMES:
Average pain score | 1 month
  Change in average pain score (NRS 0-10, 0 = painless, 10 = most painful)